CLINICAL TRIAL: NCT03463772
Title: In Vitro Maturation Versus Standard in Vitro Fertilization in Infertile Patients Diagnosed With Polycystic Ovaries Syndrome: a Study Protocol for a Single-center Prospective, Randomized Controlled Clinical Trial
Brief Title: IVM Versus Standard IVF in Infertile Patients Diagnosed With PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jie Qiao (Other)
Responsible Party: Sponsor-Investigator, Jie Qiao, President, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVM/IVF-PCOS
Record Dates: First submitted 2018-01-29; First posted 2018-03-13 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: PCOS
Keywords: in vitro maturation; polycystic ovarian syndrome; oocyte
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — In Vitro Oocyte Maturation Techniques

STUDY DESIGN:
Intervention Model Description: Eligible patients that have provided informed consent will be randomized to either IVM or standard IVF. Randomization and allocation of patients to study groups will be performed on the day 2 or 3 of the menstrual cycle. Randomization will be centrally controlled by administrative staff in the trial center, who are not involved in the treatment procedure. When there is an eligible participant to be enrolled into the study, nurses from the specific site will log in the trial center to get allocation of patients according to a computer-generated randomization list in a 1:1 ratio, with a variable block size of 2, 4 or 8 and stratified by center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard IVF (Active Comparator): On the Day2/3 of the menstrual cycle, qualified participants will be randomized into either of two groups. Participants in group A will receive standard IVF procedure. Other standard assisted reproductive treatments are similar and parallel between two groups.
  Interventions: Procedure: standard IVF
- In vitro maturation (Active Comparator): On the Day2/3 of the menstrual cycle, qualified participants will be randomized into either of two groups. Participants in group B will receive IVM procedure.Other standard assisted reproductive treatments are similar and parallel between two groups.
  Interventions: Drug: In vitro maturation

INTERVENTIONS:
Procedure: standard IVF — Ovarian stimulation will be performed by a standard protocol using gonadotrophin-releasing hormone antagonist (GnRH-ant) in association with recombinant FSH (rFSH) and human chorionic gonadotrophin (hCG).Oocyte retrieval is scheduled for 36 (±2) after hCG injection.The retrieved cumulus oocyte complexes (COC) will be inseminated using ICSI or conventional IVF according to the seman analysis. All embryos will be cultured to blastocyst stage and be vitrified.
  Arms: standard IVF
Drug: In vitro maturation — Controlled ovarian stimulation protocol will not performed in this group patients. Transvaginal ultrasound scanning was examined on natural cycle to monitor the follicle size in group B participants. Oocyte retrieval was scheduled once the endometrium had reached at least 6 mm in thickness and there was no follicle larger than 10 mm. After oocyte retrieval, the COCs will be cultured for 28-32h in special IVM media in order to get the matured oocytes. All the metaphase II (MII) oocytes were inseminated by means of intracytoplasmic sperm injection (ICSI). All embryos will be cultured to blastocyst stage and be vitrified.
  Other Names: IVM
  Arms: In vitro maturation

SUMMARY:
A single center, prospective, open-label, non-inferiority randomized controlled clinical trials (1:1 treatment ratio) regarding pregnancy outcomes between IVM and standard IVF among infertility couples with PCOS in China.

DETAILED DESCRIPTION:
A single center, randomized controlled clinical trial will enroll 350 couples with PCOS undergoing their first cycle of IVF. The participation in this study will be approximately 2 years with a total of 7 visits from the cycle beginning, pregnancy to delivery. On day 2 or day 3 following the onset of menstrual bleeding, eligible patients will be allocated to two groups at a ratio of 1:1- IVM protocol, and standard IVF protocol. All participants will be randomized through stratified block randomization according to the study sites.

ELIGIBILITY:
Inclusion Criteria:

1. Infertile couples scheduled for their first IVF cycle.
2. Women diagonosed with polycystic ovarian syndrome.
3. Voluntary participation and informed consent obtained.

Exclusion Criteria:

1. Couple with contraindication for IVF or ICSI.
2. Couples receiving donor sperm or donor eggs.
3. Couples with indications or have plan to receive PGD and PGS.
4. Sperm analysis diagnosed as azoospermia;
5. Either male partner or female partner with an abnormal chromosome karyotype (chromosome polymorphisms was not included).
6. Women who have undergone unilateral ovariectomy.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
the proportion of ongoing pregnancy leading to live birth | after 22 weeks of gestation
  number of ongoing pregnancy leading to live birth resulting from the first oocyte retrieval cycle after the randomization ( 6 month) divided by the number of patients with oocyte retrieval

SECONDARY OUTCOMES:
implantation | 28 days after embryo transfer
  Number of gestational sacs observed per embryo transferred
clinical pregnancy | 7 weeks after embryo transfer
  one or more observed gestational sac or definitive clinical signs of pregnancy under ultrasonography at 7 weeks after embryo transfer (including clinical documented ectopic pregnancy)
Miscarriage | 28 weeks of gestation
  Spontaneous loss of an intra-uterine pregnancy prior to 28 completed weeks of gestational age
Preterm birth | 28-37 weeks of pregnancy
  Birth of a fetus delieved after 28 and before 37 completed weeks of gestational age in participants confirmed ongoing pregnancy
Birth weight | within 2 weeks after live birth
  Including low birth weight (defined as weight <2500 gm at birth), very low birth weight (defined as < 1500 gm at birth), high birth weight (defined as > 4000 gm at birth) and very high birth weight (defined as > 4500 gm at birth).
Large for gestational age | within 2 weeks after live birth
  Birth weight >90th centile for gestation, based on standardised ethnicity based charts.
Small for gestational age | within 2 weeks after live birth
  Less than 10th centile for gestational age at delivery based on standardised ethnicity based charts.
Congenital anomaly | within 2 weeks after live birth
  Any congenital anomaly will be included diagnosed by physical examinition, ultrasound or necessary testing (including CT, X-ray etc.)
Perinatal mortality | within 2 weeks after live birth
  Fetal or neonatal death occurring during late pregnancy (at 28 completed weeks of gestational age and later), during childbirth, or up to seven completed days after birth.
Moderate/severe ovarian hyperstimulation syndrome (OHSS) | From date of controlled ovarian hyperstimulation until the date of oocyte retrieval, assesses about 14-16 days.
  exaggerated systemic response to ovarian stimulation characterized by a wide spectrum of clinical and laboratory manifestations. It is classified as mild, moderate, or severe according to the degree of abdominal distention, ovarian enlargement and respiratory hemodynamic, and metabolic complications. Diagosised by ultrasound, blood testing and physical examination according the Chinese Medical Guildline.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiao, Study Director — Peking University Third Hospital
Locations (1):
- Peking University third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zheng X, Guo W, Zeng L, Zheng D, Yang S, Xu Y, Wang L, Wang R, Mol BW, Li R, Qiao J. In vitro maturation without gonadotropins versus in vitro fertilization with hyperstimulation in women with polycystic ovary syndrome: a non-inferiority randomized controlled trial. Hum Reprod. 2022 Jan 28;37(2):242-253. doi: 10.1093/humrep/deab243. PMID 34849920
- [Derived] Zheng X, Guo W, Zeng L, Zheng D, Yang S, Wang L, Wang R, Mol BW, Li R, Qiao J. Live birth after in vitro maturation versus standard in vitro fertilisation for women with polycystic ovary syndrome: protocol for a non-inferiority randomised clinical trial. BMJ Open. 2020 Apr 14;10(4):e035334. doi: 10.1136/bmjopen-2019-035334. PMID 32295778